CLINICAL TRIAL: NCT01697007
Title: A Phase II Trial to Assess the Safety and Immunogenicity of DNA Priming Administered by the ID Zetajet® With or Without ID Derma Vax™ Electroporation Followed by IM MVA Boosting in Healthy Volunteers in Tanzania and Mozambique
Acronym: TaMoVac II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Collaborators: Swedish Institute for Infectious Disease Control (Other); Karolinska Institutet (Other); US Military HIV Research Program (Network); Medical Research Council (Other Government); National Institute for Medical Research, Tanzania (Other Government); Ludwig-Maximilians - University of Munich (Other); Imperial College London (Other); Mbeya medical research program (Unknown); Instituto Nacional de Saúde, Mozambique (Other Government)
Responsible Party: Principal Investigator, Patricia Jane Munseri, Prof Eligius Lyamuya, Muhimbili University of Health and Allied Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: TaMoVac II
Record Dates: First submitted 2012-09-22; First posted 2012-10-02 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Vaccines; HIV; Safety; Immunogenicity
MeSH Terms: interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 injections of DNA administered by Zetajet (Experimental): This arm will receive 600 micrograms of HIVIS DNA given as 2 injections using the Zetajet device each injection will comprise of 0.1 ml at a concentration of 3mg/ml
  Interventions: Biological: HIVIS DNA vaccine; Device: Zetajet; Biological: Modified Vaccinia Ankara (MVA-CDMR)
- 2 injections DNA by Zetajet and electroporation (Experimental): This arm will receive 600 micrograms of HIVIS DNA given as 2 injections using the Zetajet device each injection will comprise of 0.1 ml at a concentration of 3mg/ml followed by electroporation using the Derma Vax device.
  Interventions: Biological: HIVIS DNA vaccine; Device: Zetajet; Device: Derma Vax Electroporation; Biological: Modified Vaccinia Ankara (MVA-CDMR)
- 1 injection DNA by Zetajet and electroporation (Experimental): This arm will receive 600 micrograms of HIVIS DNA given in 1 injection using the Zetajet device the injection will comprise of 0.1 ml at a concentration of 6mg/ml followed by electroporation using the Derma Vax device.
  Interventions: Biological: HIVIS DNA vaccine; Device: Zetajet; Device: Derma Vax Electroporation; Biological: Modified Vaccinia Ankara (MVA-CDMR)

INTERVENTIONS:
Biological: HIVIS DNA vaccine
Device: Zetajet
Device: Derma Vax Electroporation
  Arms: 1 injection DNA by Zetajet and electroporation; 2 injections DNA by Zetajet and electroporation
Biological: Modified Vaccinia Ankara (MVA-CDMR)

SUMMARY:
Electroporation will increase the efficiency of DNA priming in terms of immune responses and will lead to a dose sparing DNA vaccine regimen. Furthermore increased DNA vaccine concentration will reduce the number of shots necessary to deliver the full dose and induce comparable immune responses as with lower DNA vaccine concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Willing to undergo counselling and HIV testing.
* Have a negative antigen/antibody ELISA for HIV infection.
* Able to give informed consent.
* Basic abilities to read and write.
* Satisfactory completion of an assessment of understanding prior to enrolment defined as 90% correct answers after three opportunities to take test.
* Resident of the region where the study is taking place.
* At low risk of HIV infection.
* Verbal assurances for adequate birth control measures.
* Healthy as evidenced by clinical and laboratory measures

Exclusion Criteria:

* At risk of HIV infection.
* Active tuberculosis.
* A history of immunodeficiency, ongoing medical and/or psychiatric condition and/or chronic illness requiring continuous or frequent medical intervention.
* Autoimmune disease.
* Hives and severe eczema.
* Substance abuse problems.
* History of grand-mal epilepsy.
* Received blood or blood products or immunoglobulins in the past 3 months.
* Receiving immunosuppressive therapy such as systemic corticosteroids or cancer chemotherapy.
* Use of experimental therapeutic agents within 30 days of study entry.
* History of cardiac disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The presence of an interferon gamma ELISpot responses to a pool of HIV peptides encoded by the vaccine to which there was no response at baseline | 2 weeks after the last vaccination
Grade 3 or above local and systemic solicited adverse events | Within 2 weeks post each immunization up to week 64 from enrollment

SECONDARY OUTCOMES:
The presence of CD4+ and CD8+ T-cell cytokine responses to pools of HIV peptides assessed by Intracellular cytokine staining | 2 weeks post last vaccination

OTHER OUTCOMES:
Any grade of adverse event that results in a clinical decision to discontinue further immunizations. | After receiving the first immunization until 64 weeks from enrollment
The presence of HIV-specific binding antibodies and the titer when these are present | Up to week 64 from enrollment
The presence of neutralizing antibodies and the titer when these are present | Approximately between week 64-68 after enrollment
The magnitude of interferon gamma ELISpot responses measured by the number of spot forming cells per million PBMCs in response to pools of HIV-peptides in the assay | 2 weeks post the last vaccination
Any grade of adverse event that occurs in a participant that has received at lease one immunization | After the first immunization up to 64 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Instituto Nacional de Saude, Maputo, Mozambique
- Tanzania (2):
  - Muhimbili University of Health and Allied Sciences, Dar es Salaam
  - Mbeya Medical Research Programme, Mbeya

REFERENCES:
- [Derived] Chissumba RM, Luciano A, Namalango E, Bauer A, Bhatt N, Wahren B, Nilsson C, Geldmacher C, Scarlatti G, Jani I, Kestens L; TaMoVac II group. Regulatory T cell abundance and activation status before and after priming with HIVIS-DNA and boosting with MVA-HIV/rgp140/GLA-AF may impact the magnitude of the vaccine-induced immune responses. Immunobiology. 2018 Dec;223(12):792-801. doi: 10.1016/j.imbio.2018.08.006. Epub 2018 Aug 12. PMID 30121146